CLINICAL TRIAL: NCT03631056
Title: Individual Patient Expanded Access for Acellular Tissue Engineered Vessel (ATEV) for Vascular System Injuries
Status: Approved for marketing | Type: Expanded Access
Sponsor: Humacyte, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-EA-IP
Record Dates: First submitted 2018-08-10; First posted 2018-08-15 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Vascular System Injuries
MeSH Terms: conditions — Vascular System Injuries

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Acellular Tissue Engineered Vessel (ATEV) / Human Acellular Vessel (HAV)

SUMMARY:
Individual patient expanded access requests may be considered for patients who have no other treatment options and are not eligible for an ATEV clinical study

DETAILED DESCRIPTION:
Procedure for Requesting Expanded Access:

The treating physician requesting expanded access must contact Humacyte directly with the basis for the request. Please include your contact information so that Humacyte may follow up with you directly.

General Criteria:

We will evaluate and respond to each expanded-access request that we receive on a case-by-case basis. Humacyte will consider the nature of the request, the patient's health, the available medical and scientific information about the investigational product, the balance of risk and potential benefit to the patient, the availability of investigational product, and the potential regulatory impact.

Anticipated Timing:

If you contact Humacyte as described above, Humacyte anticipates that we will acknowledge receipt within ten (10) business days or less.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult